CLINICAL TRIAL: NCT01371773
Title: Repositioning Method for Left-sided Double Lumen Tubes Introduced Into Right Mainstem Bronchus
Brief Title: Repositioning Method for Left-sided Double Lumen Tubes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Jae-Hyon Bahk, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JHBAhk_headrot
Record Dates: First submitted 2011-05-31; First posted 2011-06-13 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Airway Morbidity; Intubation Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Left-sided double lumen tube (Experimental)
  Interventions: Procedure: repositioning method for left-sided double lumen tubes

INTERVENTIONS:
Procedure: repositioning method for left-sided double lumen tubes — When a left-sided double lumen tube were placed in right mainstem bronchus, after withdrawing the tube into mid-trachea, it was re-advanced with patient's head turned right and counterclockwise rotation of the tube.

SUMMARY:
The purpose of this study is to devise repositioning method of a left-sided double lumen tube into left mainstem bronchus in case of misplacement into right mainstem bronchus.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing thoracic surgery that requires the placement of left-sided double lumen tubes

Exclusion Criteria:

* intraluminal lesion of left bronchus
* very distorted anatomy of tracheobronchial tree

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
repositioning success rate | up to 10 minutes

SECONDARY OUTCOMES:
anatomic parameters | up to 1 hours
  tracheal diameter, position of carina, angle between trachea and left mainstem bronchus

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Seo JH, Bae JY, Kim HJ, Hong DM, Jeon Y, Bahk JH. Misplacement of left-sided double-lumen tubes into the right mainstem bronchus: incidence, risk factors and blind repositioning techniques. BMC Anesthesiol. 2015 Oct 28;15:157. doi: 10.1186/s12871-015-0138-1. PMID 26511934